CLINICAL TRIAL: NCT06520579
Title: Pilot Proof of Concept, Prospective Cohort, Single-Center Study on the Effects of Behavioral Intervention on Swallowing and Voice Outcomes After Anterior Cervical Discectomy and Fusion (ACDF) Surgery
Brief Title: Anterior Cervical Discectomy and Fusion (ACDF) - Behavioral Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-00667
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Behavioral Intervention coupled with protein supplementation (Experimental): Patients will receive the behavioral intervention program comprised of hydration counseling, protein supplementation, and daily pharyngeal/laryngeal exercise for a total of 7 weeks.
  Interventions: Behavioral: Proactive pharyngeal-laryngeal Exercise Program; Dietary Supplement: Premier Protein Clear ® High Protein; Behavioral: Hydration Counseling
- Historical Control Group (No Intervention): Historical control data from subjects who underwent Anterior Cervical Discectomy and Fusion (ACDF) surgery but did not receive any behavioral intervention.

INTERVENTIONS:
Behavioral: Proactive pharyngeal-laryngeal Exercise Program — This program consists of daily proactive pharyngeal-laryngeal exercises and weekly sessions with a speech-language pathologist post surgery. One week prior to surgery participants will begin daily proactive pharyngeal-laryngeal exercises and continue these daily exercises for 6 weeks post surgery. Beginning approximately one week after surgery, participants will meet with the speech-language pathologist. Sessions will occur weekly, for approximately 6 weeks, and will last approximately 45 minutes.
  Arms: Proactive Behavioral Intervention coupled with protein supplementation
Dietary Supplement: Premier Protein Clear ® High Protein — Premier Protein Clear ® High Protein (20 grams of protein and 90 calories per 16.9 oz. drink) 1 drink daily for 7 weeks.
  Arms: Proactive Behavioral Intervention coupled with protein supplementation
Behavioral: Hydration Counseling — Daily hydration goals are based on recommended guidelines for adults, by gender, from The United States National Academy of Medicine (US NAM) and the European Food Safety Authority (ESFA) (~2.0 L/day for women; ~2.5 L/day for men of fluid intake, accounting for 20% daily fluid intake from food sources). Patients will be required to track via paper log whether they met their hydration goals daily.
  Arms: Proactive Behavioral Intervention coupled with protein supplementation

SUMMARY:
This study will prospectively recruit and enroll patients undergoing primary Anterior Cervical Discectomy and Fusion (ACDF) surgeries at NYU Langone. Participants will undergo pre-operative and six-week post-operative swallowing assessment using videofluoroscopy (VFSS). Acoustic voice samples and Patient Reported Outcome Measures (PROMs) for swallowing and voice will also be collected. Beginning one-week before surgery participants will begin a behavioral health program that will be continued for six-weeks after surgery. The primary goal of this study will be to determine whether a preventative behavioral health program improves instrumental measures of swallowing and voice six-weeks after ACDF surgery. .

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign consent form to participate in the study.
2. Age between 21- 99 years.
3. Scheduled to undergo ACDF surgery with surgeons in the departments of Neurosurgery or Orthopedic Surgery at NYU Langone.

Exclusion Criteria:

1. Patients with non-degenerative spine conditions, such as trauma, tumors, infection, radiation, and diabetes.
2. Patients with prior posterior-approach cervical spine procedures.
3. Patients undergoing ACDF revision procedures.
4. Patients who report a pre-existing dysphagia as the result of a neurological deficit or disorder, head and neck cancer treatment, and/or muscular condition.
5. Pregnancy. Female subjects must confirm they are not pregnant before enrolling in the study.
6. Patients with chronic kidney disease, limiting their ability to consume high levels of protein.
7. Patients with known allergies to ingredients listed in Premier Protein Clear drinks.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in pharyngeal constriction | Baseline, 6 weeks post-op
  Outcome measure will be assessed using 2D lateral videofluoroscopic images will be used to measure pharyngeal constriction pre and post intervention
Change in pharyngeal shortening | Baseline, 6 weeks post-op
  Outcome measure will be assessed using 2D lateral videofluoroscopic images will be used to measure pharyngeal shortening pre and post intervention
Change in Dysphagia Score measured by The Hospital for Special Surgery Dysphagia and Dysphonia Inventory (HSS-DDI) | Baseline, 6 weeks post-op
  The HSS-DDI consists of 31 patient-reported questions to assess Dysphagia and Dysphonia. Of the 31 questions, 20 ask about swallowing using a 5-point scoring method (1-5). Scores range from 20-100, where lower scores indicate dysphagia.

SECONDARY OUTCOMES:
Change in Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) Ratings | Baseline, 6 weeks post-op
  Complete acoustic sound files will be blindly rated using the Consensus for Auditory Perceptual Evaluation of Voice (CAPE-V), a validated quantitative rating tool used for perceptual analysis of voice. It is intended to describe the severity of various auditory attributes of a voice problem. The CAPE-V is a visual analog scale that numerically rates various vocal qualities along a continuum from 0-100 based on what the experienced listener hears, with higher values indicating worse severity.
Change in Dysphonia Score measured by The Hospital for Special Surgery Dysphagia and Dysphonia Inventory (HSS-DDI) | Baseline, 6 weeks post-op
  The HSS-DDI consists of 31 patient-reported questions to assess Dysphagia and Dysphonia. Of the 31 questions, 11 ask about speaking functions using a 5-point scoring method (1-5). Scores range from 11-55, where lower scores indicate dysphonia.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Molfenter, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: smm16@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to smm16@nyu.edu. To gain access, data requestors will need to sign a data access agreement.